CLINICAL TRIAL: NCT00741039
Title: Phase II Prospective Trial of Vaccine Responses Against Pneumococcus and Influenza in Adult Cancer Patients 65 Years of Age and Older
Brief Title: Prospective Trial of Vaccine Responses Against Pneumococcus and Influenza in Adult Cancer Patients 65 Years of Age and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-005
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Lung Cancer; Prostate Cancer
Keywords: Breast; Lung; Prostate; Vaccine
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Pneumococcal Vaccines

ARMS (2):
- 1, (Experimental): Patients > or = to 65 years of age with a diagnosis of prostate, lung, and/or breast cancer will be immunized with the inactivated influenza vaccine (0.5 ml intramuscularly) and/or the 23 valent pneumococcal vaccine (0.5 ml subcutaneously or intramuscularly).
  Interventions: Biological: inactivated influenza vaccine and the 23- valent pneumococcal vaccine
- 2 (Experimental): MSKCC employee volunteer controls > or = to 65 years of age without a cancer diagnosis will be immunized with the inactivated influenza vaccine (0.5 ml intramuscularly) and/or PPV23 vaccine (Pneumovax), (0.5 ml subcutaneously or intramuscularly).
  Interventions: Biological: inactivated influenza vaccine and the PPV23 vaccine (Pneumovax)

INTERVENTIONS:
Biological: inactivated influenza vaccine and the 23- valent pneumococcal vaccine — Patients >65 years of age with a diagnosis of prostate, lung, and/or breast cancer will be immunized with the inactivated influenza vaccine (0.5 ml intramuscularly) and/or the 23-valent pneumococcal vaccine (0.5 ml subcutaneously or intramuscularly). Prior to vaccination, titers against influenza and pneumococcus will be measured, as will serum IgG levels and IgG subtypes. At 8-16 weeks after vaccination, post vaccine titers, CBC, lymphoid phenotype and function will be assessed.
  Arms: 1,
Biological: inactivated influenza vaccine and the PPV23 vaccine (Pneumovax) — MSKCC employee volunteer controls > or = to 65 years of age without a cancer diagnosis will be immunized with the inactivated influenza vaccine (0.5 ml intramuscularly)and/or PPV23 vaccine (Pneumovax), (0.5 ml subcutaneously or intramuscularly). Prior to vaccination, titers against influenza and pneumococcus will be measured. At approximately 8-16 weeks after vaccination, post vaccine titers will be measured again.
  Arms: 2

SUMMARY:
Infections due to influenza and pneumococcus can be very serious and cause death. Anyone can get these infections. However, some people are at greater risk from the disease, including people 65 and older, the very young, and people with special health problems such as people with certain types of cancer, heart, lung, or kidney disease, or diabetes. Influenza can cause a very serious lung infection (pneumonia) and increase the risk of stroke and heart attacks. Pneumococcal disease can lead to serious infections in the lungs (pneumonia), the blood (bacteremia), and the covering of the brain (meningitis). People with the special health problems mentioned above are even more likely to die from the disease. Although there are drugs to treat these infections, they are not always effective. This makes prevention of the disease through vaccination even more important.

This study will look at the body's response to influenza and pneumococcal vaccination. We want to see how well they it will protect. Immunization is the same as vaccination. Our goal is to protect as much as we can. We are doing the study because more information is needed to see how well older patients with cancer respond to these vaccines and how well they protect against disease caused by influenza and pneumococcus.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be > or = to 65 years of age.
* Patient may be an in patient or an out-patient.
* Patient must have a diagnosis of prostate, lung, or breast cancer.
* Patient must have a life expectancy of > or = to 6 months.
* Patient must have a Karnofsky score of >40%
* Patient must be willing to return to the hospital in 8-12 weeks following immunization for blood work.
* Patients must have a platelet count of >75,000 for intramuscular injection.
* Patient may be of either gender and of any ethnic background.
* Patients must be able to understand the nature and risk of the proposed study and be able to sign consent.

Volunteer eligibility:

* MSKCC employee
* Age > or = to 65 years of age
* No previous diagnosis of cancer except basal cell carcinoma, resected Stage I melanoma or in situ cervical carcinoma. Volunteers may have had a prior history of other cancers > 3 years which required only local resection, local radiation and/or hormonal therapy such as androgen blockade.
* Patients must be able to understand the nature and risk of the proposed study and be able to sign consent.

Exclusion Criteria:

* Karnofsky score <40%:
* Patients who have received an autologous or allogeneic HCT
* Active uncontrolled bacterial or fungal infection
* Hypersensitivity to egg protein (eggs or egg products), chicken proteins, or any component in the influenza vaccine
* Prior history of any life-threatening reaction after previous administration of any influenza vaccine or any component such as thimerosal (inclusion of thimerosal varies among packaging)
* Latex allergy if going to receive the influenza vaccine
* On-going neurologic disorder (mental status change, uncontrolled seizures, encephalopathy)
* Treatment or planned treatment with cyclophosphamide, ifosphamide, or > or = to 1 mg/kg prednisone or its equivalent 12 weeks within 12 weeks of vaccination.
* HIV-1,2 seropositive patients.
* Patients not signing informed consent.
* Patients receiving the seasonal influenza vaccine may not have had it within 6 months of enrollment

Healthy controls exclusion:

* Volunteers ineligible to receive either vaccine
* Volunteers unwilling or unable to sign consent
* Hypersensitivity to egg protein (eggs or egg products), chicken proteins, or any component in the influenza vaccine
* Latex allergy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trudy Small, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Cancer Patients 65 Years of Age and Older: Vaccine Responses Against Pneumococcus and Influenza in Adult Cancer Patients 65 Years of Age and Older
- Healthy Volunteers: Vaccine Responses Against Pneumococcus and Influenza in Adults 65 Years of Age and Older
Period: Overall Study
Arm/Group | Adult Cancer Patients 65 Years of Age and Older | Healthy Volunteers
Started | 102 | 25
Completed | 100 | 25
Not Completed | 2 | 0
Not completed — Patient non-compliance | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Cancer Patients 65 Years of Age and Older | Healthy Volunteers | Total
Number analyzed (Participants) | 102 | 25 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 99 | 25 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 13 | 73
  Male | 42 | 12 | 54

OUTCOME MEASURES:

1. Primary Outcome: Determine Response Rate of Patients > or = to 65 Yrs Diagnosed
Description: For Pneumovax, complete response will be either seroconversion or a >3 fold rise in titer against at least 5 of the following serotypes contained in Pneumovax (serotypes 4, 14, 19, 23, 6B, 18C, and 9V).
Time Frame: 8-16 weeks following vaccination.
Measure: Number; unit: participants
Arm/Group | Adult Cancer Patients 65 Years of Age and Older | Healthy Volunteers
Number analyzed (Participants) | 100 | 25
participants | 63 | 24

ADVERSE EVENTS:
Arm/Group | Adult Cancer Patients 65 Years of Age and Older | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/25
Other Adverse Events (participants affected / at risk) | 0/95 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes